CLINICAL TRIAL: NCT04399473
Title: Mediators and Moderators of Pain Neuroscience Education on Disability of Patients With Nonspecific Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 133302
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2022-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Usual PT Care
- Experimental group: PNE + Usual PT Care: Participants in this arm will receive PNE education in addition to Usual PT Care
  Interventions: Behavioral: Pain Neuroscience Education (PNE)

INTERVENTIONS:
Behavioral: Pain Neuroscience Education (PNE) — Participates in the experimental group will receive 15mins X 4 sessions of pain education by the eligible trained physical therapist in addition to usual care PT treatment.
  Groups: Experimental group: PNE + Usual PT Care

SUMMARY:
The purpose of this observational study is understanding the underlying mechanisms of how PNE impacts disability in chronic low back pain patients (CLBP). The investigator will explore whether the PNE effect on patient disability is mediated by changes in pain catastrophizing, pain self-efficacy and patient beliefs about pain. Also, the investigator will explore whether the effect of PNE on disability is moderated by patient expectation.The observational multisite pre-post cohort study will be conducted in PT clinics in the Kingdom of Saudi Arabia (KSA).

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the most disabling conditions and has major socio-economic consequences. The prevalence of LBP among the population worldwide ranges between 15 and 45%. In the Kingdom of Saudi Arabia (KSA), the prevalence of LBP reported being around 18.8% among the population. Patient beliefs about back pain, pain self-efficacy, pain catastrophizing and expectation all seem to play a role in recovery. In fact, clinical guidelines recommended the treatment of non-specific chronic LBP should be considered within a multi-factorial biopsychosocial (BPS) framework. Exactly how this treatment should be delivered is not clear.

Pain neuroscience education (PNE) is a cognitive-based education that helps to educate patients about pain by focusing on neurobiology, neurophysiology and the processing and representation of pain. Even though PNE as intervention helps to improve pain, disability and other patient outcome, mixed results on its efficacy have seen in many studies. Since any complicated interventions are usually assessed by their effects on outcomes such as disability and pain, most do not target these outcomes directly; instead, they target mediating factors that are assumed to cause changes in these outcomes. In particular self-efficacy, pain catastrophizing and a patient's beliefs about back pain are thought to mediate the PNE-disability relationship since most of these cognitive factors are either highly correlated with disability or predictors for disability. The justifications for choosing these potential mediating factors: (1) self-efficacy has been shown to mediate the development of disability and is the most commonly identified mediator for psychological and behavior change interventions; (2) a study has shown that higher levels of pain catastrophizing are strongly correlated with higher levels of pain intensity and disability; and (3) a study has shown that beliefs about the consequences of LBP can influence patients' perceived pain and disability. However, the mechanisms underlying PNE effects, or the effect of PNE on mediating factors and its subsequent effect on disability as an outcome, has not been yet investigated. That leads to a knowledge gap in the evidence for understanding how PNE exerts its effect on disability. Also, identifying potential moderating factors that influence the PNE-disability relationship needs further investigation. In particular, expectation is thought to moderate the PNE-disability relationship because there are studies identified a link between expectation and clinical outcomes in patients with LBP. No study has explored the relationship between expectancy and clinical outcomes in the context of PNE. So, the influence of patient expectation on the magnitude of PNE effect on disability needs investigation.

The purpose of this 18-months project is understanding the underlying mechanisms of how PNE impacts disability. This project is significant because it will help us understand how PNE works by studying the underlying mechanisms and for whom and under what circumstances will PNE produces the greatest clinical benefits on the disability for patients with chronic LBP. Knowing how certain factors work will help PTs to enhance the elements of PNE that hopefully will target patient-specific factors and subsequently will reduce disability.

ELIGIBILITY:
Inclusion Criteria:

1. Pain between the 12th rib and buttocks with or without symptoms into one or both legs which originate from the lumber region.
2. Pain >12 weeks.
3. Oswestry disability score =>20%.

Exclusion Criteria:

1. No surgery to the lumbosacral spine in the last 12 months.
2. No evidence of "Red flags" conditions (e.g., cauda equina, neurological deficits, cancer, fracture or infection).
3. Not currently receiving any intervention for LBP from other healthcare provider (e.g., physical therapy, massage therapy, etc.).
4. Not currently known to be pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Nonspecific Chronic Low Back Pain (NCLBP)
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2020-11-29 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI)(Arabic version). | 2 week.
  Change score of disability scores from baseline.

OTHER OUTCOMES:
Pain Self-Efficacy (PSE). | 2 week.
  Measured by Pain Self-efficacy Questionnaire (PSE) (Arabic version).
Pain Catastrophism. | 2 week.
  Measured by Pain Catastrophizing Scale (PCS) (Arabic version).
Patient Back Beliefs. | 2 week.
  Measured by Back Beliefs Questionnaire (BBQ) (Arabic version)
Patient Expectation. | Baseline
  Measured by short form of EXPECT Questionnaire (Arabic version).

CONTACTS AND LOCATIONS:
Locations (6):
- Saudi Arabia (6):
  - East Jeddah General Hospital-Physical Therapy Department, Jeddah, Mecca Region
  - King Abdulaziz Hospital-Rehabilitation Center, Jeddah, Mecca Region
  - King Fahad General Hospital-Physical Therapy Department, Jeddah, Mecca Region
  - King Abdullah Complex-Physical Therapy Department, Jeddah, Mecca Region
  - King Fiasal Hospital-Physical Therapy Department, Ta'if, Mecca Region
  - King Abdulaziz Hospital-Phyiscal Therapy Department, Ta'if, Mecca Region

IPD SHARING:
Plan to Share IPD: No